CLINICAL TRIAL: NCT05511467
Title: Neural Circuitries of Motor Learning as a Target to Modulate Sensorimotor Recovery After Stroke
Brief Title: Learning in Stroke
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Other Study IDs: 00116626; 5P20GM109040-10 (NIH)
Record Dates: First submitted 2022-08-09; First posted 2022-08-23 (Actual); Results first posted 2025-09-04 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Stroke; Sensorimotor Impairment
Keywords: procedural learning; maladaptive plasticity
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- stroke group
  Interventions: Behavioral: Visuomotor learning task
- control group
  Interventions: Behavioral: Visuomotor learning task

INTERVENTIONS:
Behavioral: Visuomotor learning task — Participants undergo functional magnetic resonance imaging during the performance of the visuomotor learning task. The visuomotor learning task involves holding a device in the hand that measures the strength of the grip when squeezing the 'gripper'.

SUMMARY:
After a stroke, plasticity occurs in the brain from microscopic to network level with positive but also negative consequences for functional recovery. Why post-stroke plasticity takes a beneficial or a maladaptive direction is still incompletely understood. Because the biological mechanisms underlying sensorimotor learning parallel those observed during recovery, learning mechanisms could be potential modifiers of post-stroke neuroplasticity and have a discrete mal-/adaptive impact on the recovery of sensorimotor function. This project seeks to further the understanding of the link between brain circuits that control the integration of new information during procedural learning in the injured brain and those circuits that are involved in adaptive plastic changes during recovery of sensorimotor function post-stroke. The project's methodological approach will allow the characterization of procedural learning-related neural network dynamics based on functional magnetic resonance imaging (MRI) in human volunteers with and without neurologically impairment post-stroke. Through multivariate integration of behavioral and biological descriptors of sensorimotor recovery, the project will investigate the association between motor learning-related network dynamics and descriptors of recovery.

ELIGIBILITY:
INCLUSION CRITERIA

For all participants:

* adult volunteers (age ≥18 years)
* right-hand dominance as defined by the Edinburgh Handedness Inventory

Stroke-specific inclusion criteria:

* ischemic or hemorrhagic lesion
* subcortical or cortical tissue involvement
* chronic phase (>6 months) after their index lesion
* voluntary whole-hand grip force (MRC, Medical Research Council scale for muscle force ≥2)
* repeated release (standardized as a reduction of 50% of maximum voluntary contraction measured with a dynamometer)

EXCLUSION CRITERIA

For all participants:

* Presence of any MRI risk factors
* substance use disorder
* psychotic disorders

Stroke-group specific exclusion criteria:

* Primary intracerebral hematoma
* subarachnoid hemorrhage
* bi-hemispheric or cerebellar strokes
* other concomitant neurological disorders affecting upper extremity motor function
* documented history of dementia before or after stroke
* severe aphasia, particularly of receptive nature (NIHSS Language subsection ≥2), affecting their ability to understand the purpose of the study and give informed consent
* uncontrolled hypertension despite treatment
* intake of tricyclic anti-depressants or neuroleptic medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke survivors (>6 months) after their index lesion, ≥18 years of age. Healthy adults (≥18 years of age).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2025-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period 09/01/2022 - 03/30/2024
Period: Overall Study
Arm/Group | stroke group | control group
Started | 25 | 15
Completed | 24 | 15
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | stroke group | control group | Total
Number analyzed (Participants) | 25 | 15 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 8 | 24
  >=65 years | 9 | 7 | 16
Age, Continuous [Median (Full Range); unit: years] | 59 [34 to 77] | 60 [34 to 77] | 59.5 [34 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 14 | 7 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 12 | 2 | 14
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25 | 15 | 40

OUTCOME MEASURES:

1. Primary Outcome: Learning Rate as Indexed by Change in the Precision of Visuomotor Grip Force Adjustment (i.e., Reduction of Precision Error in Force Adjustment)
Description: Isometric whole-hand grip force is captured continuously with grip-force transducers (at 1000Hz) and adjusted relative to the individual maximum voluntary contraction.
  Precision of force adjustment is based on the recorded muscle force monitored during task performance and defined as the actual force exerted by the participant relative to the target force (measurement unit: precision in %), with positive values indicating over- and negative values indicating undershoot. Learning rate from before to after learning will be defined as the difference in precision between before as compared to after one single learning session. Precision error was calculated as the percentage deviation of the actual grip force from the target force, averaged across trials before and after the learning task. A reduction in force error indexes a behavioral advantage of force adjustment over time and is thus interpreted as learning.
Time Frame: Pre Learning Session and Post Learning Session (approximately 90 minutes)
Population: One stroke group participant was excluded because of poor data quality (excessive movement inside the MRI). One control group participant excluded due to incidental findings.
Measure: Median (Full Range); unit: Percentage deviation from target force
Arm/Group | stroke group | control group
Number analyzed (Participants) | 24 | 14
Percentage deviation from target force | -1.48 [-72.6 to 45.9] | 0.303 [-16.9 to 12.4]

2. Primary Outcome: Change in Blood-oxygen-level-dependent (BOLD) Signal Derived Multi-voxel Brain Activation
Description: Learning-related BOLD-signal-derived brain activation relative to motor performance.
Time Frame: Pre Learning Session and Post Learning Session (approximately 90 minutes)
Population: as for outcome 1
Measure: Mean (90% Confidence Interval); unit: percentage of BOLD signal change
Arm/Group | stroke group | control group
Number analyzed (Participants) | 24 | 14
percentage of BOLD signal change | 2.6 [1.1 to 4.2] | 3.25 [1.8 to 4.75]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the experimental procedures (approximately 4 individual visits within 2 consecutive weeks).
Description: Adverse events were defined as unexpected events during experimental procedures, specifically including magnetic resonance imaging (MRI), related or unrelated to experimental procedures.
Arm/Group | stroke group | control group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/15
Other Adverse Events (participants affected / at risk) | 0/25 | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | stroke group (N=25) | control group (N=15)
Incidental finding during MRI (Nervous system disorders) | 0 (0) | 1 (1) — Incidental finding during magnetic resonance imaging

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-11-14): https://cdn.clinicaltrials.gov/large-docs/67/NCT05511467/Prot_SAP_001.pdf
  • Informed Consent Form (2021-12-23): https://cdn.clinicaltrials.gov/large-docs/67/NCT05511467/ICF_000.pdf